CLINICAL TRIAL: NCT02660827
Title: Safety Evaluation of the Hybrid Closed Loop (HCL) System in Pediatric Subjects With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 302
Record Dates: First submitted 2016-01-16; First posted 2016-01-21 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hybrid closed loop (Experimental): All subjects will be wearing the MMT-670G insulin pump, using it with the closed loop algorithm
  Interventions: Device: Insulin Pump

INTERVENTIONS:
Device: Insulin Pump — Closed Loop Algorithm
  Other Names: MMT-670G

SUMMARY:
This study is a single-arm, multi-center, Home and Hotel Clinical Investigation in pediatric subjects with type 1 diabetes on insulin pump therapy. The purpose of this study is to demonstrate that the closed loop algorithm is safe as part of the overall system, and to assess the PLGM feature in 7-13 years old subjects.

DETAILED DESCRIPTION:
The study will proceed as follows:

Run-in Period - General:

A total of up to 200 subjects (age 2-13) will be enrolled at up to 15 investigational centers (14 in the US, 1 EMEA) in order to reach 120 subjects who will complete the HCL study.

Study Period - At Home:

Following the two week run-in period using the Study Pump (670G), all subjects (age 2-13) will participate in a 3-month study period.

Study Period - Hotel Study Subjects (age 7-13) will participate in a Hotel study (6 days, 5 nights), with the remainder of the study period to be spent at home. Subjects 2-6 years of age are not required to participate in a hotel study. Instead, they will participate in an out-of-home study for 5 consecutive days, 4-6 hours per day.

Continued Access Program Subjects will be given the opportunity to extend use of their study devices for a period of up to 3 years . If subjects choose to participate in the continuation period, they will retain the study devices at the end of study period visit or receive them back in the event they have been returned to study staff already.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Subject is age 2-13 years at time of screening
2. Subject has a clinical diagnosis of type 1 diabetes for 1 year or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Subject age 2-6 years has a clinical diagnosis of type 1 diabetes for 3 months or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis

   Study-specific inclusion criteria
4. Subject must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units
5. Subjects 7-13: Subjects and their parent(s)/guardian(s) are willing to participate in an overnight visit at the end of the run-in period.
6. Subject 7-13 years of age and their parent(s)/guardian(s) are willing to participate in a hotel study for the specified duration of hotel stay.
7. Subject 2-6 years of age and their parent(s)/guardian(s) are willing to participate in an extended visit during the study period to perform Frequent Sample Testing.
8. Subject must have companion 18 years or older who will sleep in the same dwelling place every night during the study period. This requirement may be verified by subject report at screening visit.
9. Subject is willing to perform ≥ 4 finger stick blood glucose measurements daily
10. Subject is willing to perform required sensor calibrations
11. Subject is willing to wear the system continuously throughout the study
12. Subject has a Glycosylated hemoglobin (A1C) value less than 10.0% (as processed by Central Lab) at time of screening visit Note: All HbA1C blood specimens will be sent to and tested by a NGSP certified Central Laboratory. A1C testing must follow National Glycohemoglobin Standardization Program (NGSP) standards.
13. Subject has TSH in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
14. Subject 7 -13 years of age has had pump therapy for greater than 6 months prior to screening (with or without CGM experience)
15. Subject 2-6 years of age has had pump therapy for greater than 90 days prior to screening (with or without CGM experience)
16. Subjects and their parent(s)/guardian(s) are willing to upload data from the study pump; must have Internet access and a computer system that meets the requirements for uploading the study pump
17. If subject has celiac disease, it has been adequately treated as determined by the investigator
18. Subjects and their parent(s)/guardian(s) are willing to take one of the following insulins and can financially support the use of either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount)

    * Humalog® (insulin lispro injection)
    * NovoLog® (insulin aspart)
19. Subjects and their parent(s)/guardian(s)/companions must be able to speak and be literate in English as verified by the investigator

Exclusion Criteria:

1. Subject has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:

   1. Medical assistance (i.e. Paramedics, Emergency Room ( ER) or Hospitalization)
   2. Coma
   3. Seizures
2. Subject is unable to tolerate tape adhesive in the area of sensor placement
3. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
4. Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
5. Subject has a cardiovascular condition which the investigator determines should exclude the subject, i.e. ventricular rhythm disturbance, hypertrophic cardiomyopathy
6. Subject is being treated for hyperthyroidism at time of screening
7. Subject has diagnosis of adrenal insufficiency
8. Subject 7-13 years of age has had DKA in the 6 months prior to screening visit.
9. Subject 2-6 years of age has had DKA in the 3 months prior to screening visit
10. Subject has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study
11. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
12. Subject 7-13 years of age has been hospitalized or has visited the ER in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes
13. Subject 2-6 years of age has been hospitalized or has visited the ER in the 3 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes
14. Subject is currently abusing illicit drugs
15. Subject is currently abusing marijuana.
16. Subject is currently abusing prescription drugs
17. Subject is currently abusing alcohol
18. Subject is using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening
19. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
20. Subject has elective surgery planned that requires general anesthesia during the course of the study
21. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
22. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
23. Subject diagnosed with current eating disorder such as anorexia or bulimia
24. Subject has been diagnosed with chronic kidney disease that results in chronic anemia
25. Subject has a hematocrit that is below the normal reference range of lab used.
26. Subject is on dialysis
27. Subject has serum creatinine of >2 mg/dL.

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - AMCR Institute, Escondido, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - SoCal Diabetes, Torrance, California
  - Barbara Davis Center, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of South Florida - USF Health, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
- Sheba Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forlenza GP, Ekhlaspour L, DiMeglio LA, Fox LA, Rodriguez H, Shulman DI, Kaiserman KB, Liljenquist DR, Shin J, Lee SW, Buckingham BA. Glycemic outcomes of children 2-6 years of age with type 1 diabetes during the pediatric MiniMed 670G system trial. Pediatr Diabetes. 2022 May;23(3):324-329. doi: 10.1111/pedi.13312. Epub 2022 Jan 31. PMID 35001477
- [Derived] Forlenza GP, Pinhas-Hamiel O, Liljenquist DR, Shulman DI, Bailey TS, Bode BW, Wood MA, Buckingham BA, Kaiserman KB, Shin J, Huang S, Lee SW, Kaufman FR. Safety Evaluation of the MiniMed 670G System in Children 7-13 Years of Age with Type 1 Diabetes. Diabetes Technol Ther. 2019 Jan;21(1):11-19. doi: 10.1089/dia.2018.0264. Epub 2018 Dec 26. PMID 30585770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 subjects aged 2-13 years entered study period, 1 subject withdrawn during study period, 5 subjects didn't participate continued access period after finishing study period; 145 subjects aged 2-13 years entered continued access period, 25 subjects withdrawn and 120 subjects completed continued access period.
Pre-assignment Details: 2-13 years subjects wearing MMT-670G insulin pump
Groups:
- Subjects Wearing MMT-670G Insulin Pump: Subjects wearing MMT- 670G insulin pump during Study and Continued Access period
Period: From Study to End of Continued Access
Arm/Group | Subjects Wearing MMT-670G Insulin Pump
Started | 151
Completed | 120
Not Completed | 31
Not completed — Withdrawal by Subject | 21
Not completed — Withdrawal by Sponsor | 2
Not completed — Adverse Event | 3
Not completed — didn't participate continued access period | 5
Period: Period 1: Study Period
Arm/Group | Subjects Wearing MMT-670G Insulin Pump
Started | 151
Completed | 150
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 2: Continued Access Period
Arm/Group | Subjects Wearing MMT-670G Insulin Pump
Started | 145
Completed | 120
Not Completed | 25
Not completed — Withdrawal by Subject | 20
Not completed — Withdrawal by Sponsor | 2
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: 2-13 Years old subjects wearing MMT-670G insulin pump
Groups:
- Age 2-13 Yrs: Age 2-13 Yrs Subjects wearing MMT- 670G insulin pump
Arm/Group | Age 2-13 Yrs
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 132
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 140
  Israel | 11
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] — Population: One Subject's height and weight were not measured at enrollment.
  kg/m^2
    number analyzed (Participants) | 150
    (all) | 18.4 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Age 2-13 Years Old Subjects Change in A1C
Description: Descriptive analysis of change in A1C from baseline to end of 3-month study period
Time Frame: Baseline and end of 3-month study period
Population: 2-13 years old subjects wearing MMT-670G insulin pump; two subjects end of study A1C not collected.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Groups:
- Age 2-13 Years Old Wearing MMT-670G Insulin Pump: 2-13 years old subjects wearing MMT-670G insulin pump.
Arm/Group | Age 2-13 Years Old Wearing MMT-670G Insulin Pump
Number analyzed (Participants) | 149
percentage of hemoglobin | -0.37 (0.62)

2. Secondary Outcome: Age 2-13 Years Old Subjects Mean Change in % of Time in Euglycemia (70-180 mg/dL)
Description: mean change in % of time in Euglycemia (70-180 mg/dL) from baseline to 3 months study period
Time Frame: baseline and 3 months
Population: 2-13 years old subjects wearing MMT-670G insulin pump.
Measure: Mean (Standard Deviation); unit: Percentage of time
Groups:
- Age 2-13 Years Old Wearing the MMT-670G Insulin Pump: 2-13 years old subjects wearing MMT-670G insulin pump.
Arm/Group | Age 2-13 Years Old Wearing the MMT-670G Insulin Pump
Number analyzed (Participants) | 151
Percentage of time | 8.58 (8.84)

3. Secondary Outcome: Age 2-13 Years Old Subjects Mean Change in % of Time in Hyperglycemia (> 180 mg/dL)
Description: mean change in % of time in hyperglycemia (> 180 mg/dL) from baseline to 3 months study period
Time Frame: baseline and 3 months
Population: 2-13 years old subjects wearing MMT-670G insulin pump.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Age 2-13 Years Old Wearing the MMT-670G Insulin Pump
Number analyzed (Participants) | 151
Percent of time | -7.39 (9.96)

4. Secondary Outcome: Age 2-13 Years Old Subjects Mean Change in % of Time in Hypoglycemia (<70 mg/dL)
Description: mean change in % of time in hypoglycemia (< 70 mg/dL) from baseline to 3 months study period
Time Frame: baseline and 3 months
Population: 2-13 years old subjects wearing MMT-670G insulin pump.
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Age 2-13 Years Old Wearing the MMT-670G Insulin Pump
Number analyzed (Participants) | 151
percent of time | -1.19 (2.58)

5. Secondary Outcome: Age 2-13 Years Old - Number of Severe Hypoglycemic Event
Description: Number of severe hypoglycemic events occurred during 3-month study period.
Time Frame: 3 months
Population: 2-13 years old subjects wearing MMT-670G insulin pump.
Measure: Number; unit: events
Arm/Group | Age 2-13 Years Old Wearing the MMT-670G Insulin Pump
Number analyzed (Participants) | 151
events | 0

6. Secondary Outcome: Age 2-13 Years Old - Number of Diabetic Ketoacidosis (DKA) Event
Description: Number of Diabetic Ketoacidosis (DKA) events occurred during 3-month study period.
Time Frame: 3 months
Population: 2-13 years old subjects wearing MMT-670G insulin pump.
Measure: Number; unit: events
Arm/Group | Age 2-13 Years Old Wearing the MMT-670G Insulin Pump
Number analyzed (Participants) | 151
events | 0

7. Secondary Outcome: Age 7-13 Years Old Subjects PLGM Performance - Event Rate Without Hypoglycemia at YSI-FST <=65 mg/dL
Description: Event rate without Hypoglycemia at YSI-FST <=65 mg/dL among 105 subjects who underwent the PLGM experiments. The event rate without hypoglycemia is the number of experiments without hypoglycemia/total number of experiments and hypoglycemic events are defined based on the occurrence of 2 or more continuous YSI-FST <= 65mg/dL during in-clinic procedures.
Time Frame: Up to 12 hours after the start of PLGM period
Population: 7-13 years old subjects wearing MMT-670G insulin pump, participating in clinical evaluation of the suspend before low feature.
Measure: Number; unit: percentage of total experiments
Groups:
- Age 7-13 Years Old Wearing the MMT-670G Insulin Pump: 7-13 years old subjects wearing MMT-670G insulin pump, participating in clinical evaluation of the suspend before low feature.
Arm/Group | Age 7-13 Years Old Wearing the MMT-670G Insulin Pump
Number analyzed (Participants) | 105
percentage of total experiments | 84.8

ADVERSE EVENTS:
Time Frame: 3 months for Study period, up to 3 years for Continued Access period.
Groups:
- Age 2-13 Yrs Study Period: 2-13 years old subjects wearing MMT-670G insulin pump during Study period.
- Age 2-13 Yrs Continued Access Period: 2-13 years old subjects wearing MMT-670G insulin pump during Continued Access period.
Arm/Group | Age 2-13 Yrs Study Period | Age 2-13 Yrs Continued Access Period
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/151 | 4/145
Other Adverse Events (participants affected / at risk) | 88/151 | 113/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 2-13 Yrs Study Period (N=151) | Age 2-13 Yrs Continued Access Period (N=145)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 2-13 Yrs Study Period (N=151) | Age 2-13 Yrs Continued Access Period (N=145)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acetonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood ketone body increased (Investigations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 3 (3)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 4 (4)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 6 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Dacryocanaliculitis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 6 (8)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema infectiosum (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 7 (8) | 15 (17)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 6 (10)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 2 (2)
Greenstick fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Helicobacter test positive (Investigations) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 56 (146) | 70 (372)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 7 (8)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1) | 5 (5)
Injury associated with device (General disorders) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Medical device site abscess (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 2 (2) | 0 (0)
Medical device site rash (General disorders) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 8 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 5 (5)
Otitis media acute (Infections and infestations) | 0 (0) | 5 (6)
Pain (General disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Periumbilical abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 14 (15)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 7 (7)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 6 (7)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Torus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 20 (28)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 5 (5) | 8 (9)
Viral pharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02660827/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT02660827/SAP_001.pdf